CLINICAL TRIAL: NCT05889403
Title: Evaluation of the Patient's Autonomy Vis-à-vis the Therapeutic Project Proposed in a Chronic Pain Structure
Acronym: DoulEthic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DoulEthic
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patient autonomy is recognized throughout the world, by caregivers, as a value. The idea of autonomy has been the keystone of the changes accomplished in the contemporary history of health law. It is about respect for everyone to have their own health and to choose the options that correspond to their wishes, their values or their life projects. The recently revised definition of pain specifies that it is "an unpleasant sensory and emotional experience associated with, or resembling that associated with, actual or potential tissue damage". In this, pain is always a personal experience that is influenced to varying degrees by biological, psychological and social factors. The High Authority of Health considers pain as chronic is considered when it is persistent or recurrent beyond what is usual for its presumed initial cause (most often beyond 3 months), that it responds harm to treatment and that they induce a significant and progressive deterioration of functional and relational capacities. Chronic pain confines patients on a psychosocial level. It is no longer just a symptom, it is even a disease in its own right since 2019 with the new classification of diseases proposed by the World Health Organization.In France, chronic pain concerns 31.7% of French people regardless of its intensity, and 19.9% of French people for moderate to severe pain, which represents 13 million people in total. As with any chronic disease, the patient suffering from persistent pain must develop the ability to adapt to cope with the new situation with which he is confronted. He must be able to acquire knowledge and new know-how related to his pathology and thus finally find a new homeostasis, a new state of health having integrated "the pathological state". In France, chronic pain concerns 31.7% of French people regardless of its intensity, and 19.9% of French people for moderate to severe pain, which represents 13 million people in total. As with any chronic disease, the patient suffering from persistent pain must develop the ability to adapt to cope with the new situation with which he is confronted. He must be able to acquire knowledge and new know-how related to his pathology and thus finally find a new homeostasis, a new state of health having integrated "the pathological state".In France, chronic pain concerns 31.7% of French people regardless of its intensity, and 19.9% of French people for moderate to severe pain, which represents 13 million people in total. As with any chronic disease, the patient suffering from persistent pain must develop the ability to adapt to cope with the new situation with which he is confronted. He must be able to acquire knowledge and new know-how related to his pathology and thus finally find a new homeostasis, a new state of health having integrated "the pathological state".

In current practice, this skill is assessed in case of doubt (generally when there is uncertainty about the patient's understanding of the issues and his involvement in the therapeutic project) intuitively, by following a Socratic questioning or from grids like the MacCAT-T. In the pain center, investigators use the MacCAT-T but investigators have not yet systematically measured the benefit and the cost of using this questionnaire in everyday practice. In particular, investigators want to know if the skill is not overestimated by the doctor in charge of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient coming in 1st chronic pain consultation
* French-speaking patient

Exclusion Criteria:

* Patient with a significant visual or auditory deficit
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objects to the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient coming in 1st chronic pain consultation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of patient autonomy | Day 1
  This outcome corresponds to the analysis of the distribution (means, standard deviations, medians, etc.) of MacCAT-T subscores (understanding, evaluation, appreciation and reasoning) of patients just after the pain consultation, where the personalized therapeutic plan was offered to them.
  analysis of the distribution (means, standard deviations, medians, etc.) of MacCAT-T subscores (understanding, evaluation, appreciation and reasoning) of patients just after the pain consultation, where the personalized therapeutic plan was offered to them

SECONDARY OUTCOMES:
Good capacity for evaluation by the investigators of the autonomy of their patient | Day 1
  This outcome corresponds to the the percentage of concordance between the assessment (on a 3-point scale: not deficient, moderately deficient, very deficient) of the patient's degree of autonomy by the pain physician and the score obtained on the MacCAT-T.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Hôpital Saint-Joseph, Paris, France

REFERENCES:
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Bouhassira D, Lanteri-Minet M, Attal N, Laurent B, Touboul C. Prevalence of chronic pain with neuropathic characteristics in the general population. Pain. 2008 Jun;136(3):380-387. doi: 10.1016/j.pain.2007.08.013. Epub 2007 Sep 20. PMID 17888574
- [Background] Engel GL. The need for a new medical model: a challenge for biomedicine. Science. 1977 Apr 8;196(4286):129-36. doi: 10.1126/science.847460.
- [Background] Grisso T, Appelbaum PS, Hill-Fotouhi C. The MacCAT-T: a clinical tool to assess patients' capacities to make treatment decisions. Psychiatr Serv. 1997 Nov;48(11):1415-9. doi: 10.1176/ps.48.11.1415. PMID 9355168
- [Background] Raffard S, Lebrun C, Laraki Y, Capdevielle D. Validation of the French Version of the MacArthur Competence Assessment Tool for Treatment (MacCAT-T) in a French Sample of Individuals with Schizophrenia: Validation de la version francaise de l'instrument d'evaluation des competences MacArthur-traitement (MacCAT-T) dans un echantillon francais de personnes souffrant de schizophrenie. Can J Psychiatry. 2021 Apr;66(4):395-405. doi: 10.1177/0706743720966443. Epub 2020 Oct 16. PMID 33064578
- [Background] Etchells E, Darzins P, Silberfeld M, Singer PA, McKenny J, Naglie G, Katz M, Guyatt GH, Molloy DW, Strang D. Assessment of patient capacity to consent to treatment. J Gen Intern Med. 1999 Jan;14(1):27-34. doi: 10.1046/j.1525-1497.1999.00277.x. PMID 9893088